CLINICAL TRIAL: NCT03310450
Title: Predictors of Cardiac Troponin Release After Tour de Borobudur 2017
Brief Title: Tour de Borobudur Troponin Study on Predictors and Synergistic Role of MDA and Hs-CRP Levels
Acronym: TdBTS
Status: Completed | Type: Observational
Sponsor: Universitas Negeri Semarang (Other)
Collaborators: Ministry of Research, Technology and Higher Education, Republic of Indonesia (Unknown); Universitas Diponegoro (Other)
Responsible Party: Sponsor
Other Study IDs: 0017
Record Dates: First submitted 2017-10-02; First posted 2017-10-16 (Actual); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Heart Arrest; Sport Injury; Inflammatory Response; Oxidative Stress
Keywords: troponin-I; hs-CRP; Malondialdehyde; predictors
MeSH Terms: conditions — Heart Arrest | interventions — Health Records, Personal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 140kms cycling: Participants of Tour de Borobudur 2017 140 km cycling touring and willing to participate in the study.
  Investigator did not give any intervention, just observed the cycling touring event that the subjects participated
  Interventions: Other: 140kms cycling
- Group 100kms cycling: Participants of Tour de Borobudur 2017 100 km cycling touring and willing to participate in the study.
  Investigator did not give any intervention, just observed the cycling touring event that the subjects participated
  Interventions: Other: 140kms cycling
- Group 240kms cycling: Participants of North Coast 2017 240 km cycling touring and willing to participate in the study.
  Investigator did not give any intervention, just observed the cycling touring event that the subjects participated
  Interventions: Other: 140kms cycling

INTERVENTIONS:
Other: 140kms cycling — Main exposure is long distance cycling touring (TdB/NC) consists of three groups; 140kms, 100kms, and 240kms (investigator did not give any treatment/intervention, just observed the cycling touring event)
  Other Names: medical history; sports participation history; clinical appearance; lipid profile status

SUMMARY:
Prospective observational study to determine predictors that related to cardiac troponin I (cTnI) release, malondialdehyde (MDA) and high sensitivity C Reactive Protein (hs-CRP) after Tour de Borobudur (TdB) 2017

DETAILED DESCRIPTION:
Eligible Criteria:

1. minimum sample size of 80 men, non-athlete, participants of TdB
2. Classified into two groups: 160kms cycling and 100kms cycling participation
3. 25-55 years old
4. voluntary participate in the research
5. eligible in pre participatory physical examination and ECG test by the doctor
6. have no history of the previous acute coronary syndrome (ACS)

Measurements:

Interview for determining predictors of sports participation history, medical history, family medical history and Rate of Perceived Exertion Measurement and examination to determine: anthropometry parameters, clinical conditions (Systolic BP, Diastolic BP, hemoglobin levels, T-cholesterol and HDL-C levels, the intensity in cycling activities (mileage, velocity, duration, and time for resting), hemodynamic responses (average and maximum heart rate, Karvonen Index), and Hydration status

Other outcome measurements; pre and post-TdB 2017 measurements of cTnI, MDA, and hs-CRP

ELIGIBILITY:
Inclusion Criteria:

* minimum sample size of 80 men, non athlete, participants of TdB
* Classified into two groups: 160kms cycling and 100kms cycling participation
* 25-55 years old
* voluntary participate in the research
* eligible in pre participatory physical examination and ECG test by doctor have no history of previous acute coronary syndrome (ACS)

Exclusion Criteria:

* stop cycling before finish line due to mechanical or bicycle related errors
* (subjects who stop cycling due to any physical symptoms and health related problem included in analysis)

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: participants of Tour de Borobudur Indonesia 2017
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2017-10-28 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2018-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahalul Azam, Dr, Principal Investigator — Universitas Negeri Semarang
Locations (1):
- Universitas Negeri Semarang, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Serrano-Ostariz E, Terreros-Blanco JL, Legaz-Arrese A, George K, Shave R, Bocos-Terraz P, Izquierdo-Alvarez S, Bancalero JL, Echavarri JM, Quilez J, Aragones MT, Carranza-Garcia LE. The impact of exercise duration and intensity on the release of cardiac biomarkers. Scand J Med Sci Sports. 2011 Apr;21(2):244-9. doi: 10.1111/j.1600-0838.2009.01042.x. PMID 19919634
- [Background] Grande G, Romppel M, Glaesmer H, Petrowski K, Herrmann-Lingen C. The type-D scale (DS14) - Norms and prevalence of type-D personality in a population-based representative sample in Germany. Pers Individ Dif [Internet]. 2010;48(8):935-9. Available from: http://dx.doi.org/10.1016/j.paid.2010.02.026
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] Kleinbaum DG, Kupper LL, Morgenstern H. Epidemiologic research; Principles and quantitative methods. New York: John Wiley and Son Inc; 1982. 1-527 p.
- [Background] Bahrudin U, Morikawa K, Takeuchi A, Kurata Y, Miake J, Mizuta E, Adachi K, Higaki K, Yamamoto Y, Shirayoshi Y, Yoshida A, Kato M, Yamamoto K, Nanba E, Morisaki H, Morisaki T, Matsuoka S, Ninomiya H, Hisatome I. Impairment of ubiquitin-proteasome system by E334K cMyBPC modifies channel proteins, leading to electrophysiological dysfunction. J Mol Biol. 2011 Nov 4;413(4):857-78. doi: 10.1016/j.jmb.2011.09.006. Epub 2011 Sep 12. PMID 21939669
- [Background] Bahrudin U, Morisaki H, Morisaki T, Ninomiya H, Higaki K, Nanba E, Igawa O, Takashima S, Mizuta E, Miake J, Yamamoto Y, Shirayoshi Y, Kitakaze M, Carrier L, Hisatome I. Ubiquitin-proteasome system impairment caused by a missense cardiac myosin-binding protein C mutation and associated with cardiac dysfunction in hypertrophic cardiomyopathy. J Mol Biol. 2008 Dec 26;384(4):896-907. doi: 10.1016/j.jmb.2008.09.070. Epub 2008 Oct 7. PMID 18929575
- [Background] Purwowiyoto SL, Aryadi A, Suryaatmadja B, Ruray D, Purwowiyoto BS, Siswanto BB. Positive correlation between ECG dispersion mapping (heartvueTM) with T2DM patients. Glob Heart [Internet]. 2014;9(1):e243. Available from: http://linkinghub.elsevier.com/retrieve/pii/S221181601402119X
- [Background] de Koning L, Merchant AT, Pogue J, Anand SS. Waist circumference and waist-to-hip ratio as predictors of cardiovascular events: meta-regression analysis of prospective studies. Eur Heart J. 2007 Apr;28(7):850-6. doi: 10.1093/eurheartj/ehm026. Epub 2007 Apr 2. PMID 17403720
- [Background] Shave R, George KP, Atkinson G, Hart E, Middleton N, Whyte G, Gaze D, Collinson PO. Exercise-induced cardiac troponin T release: a meta-analysis. Med Sci Sports Exerc. 2007 Dec;39(12):2099-106. doi: 10.1249/mss.0b013e318153ff78. PMID 18046180
- [Background] Morrow DA. Troponins in patients with acute coronary syndromes: biologic, diagnostic, and therapeutic implications. Cardiovasc Toxicol. 2001;1(2):105-10. doi: 10.1385/ct:1:2:105. PMID 12213981
- [Background] Jassal DS, Moffat D, Krahn J, Ahmadie R, Fang T, Eschun G, Sharma S. Cardiac injury markers in non-elite marathon runners. Int J Sports Med. 2009 Feb;30(2):75-9. doi: 10.1055/s-0028-1104572. Epub 2009 Jan 28. PMID 19177312
- [Background] Rodondi N, Marques-Vidal P, Butler J, Sutton-Tyrrell K, Cornuz J, Satterfield S, Harris T, Bauer DC, Ferrucci L, Vittinghoff E, Newman AB; Health, Aging, and Body Composition Study. Markers of atherosclerosis and inflammation for prediction of coronary heart disease in older adults. Am J Epidemiol. 2010 Mar 1;171(5):540-9. doi: 10.1093/aje/kwp428. Epub 2010 Jan 28. PMID 20110287
- [Background] Eijsvogels TM, Hoogerwerf MD, Maessen MF, Seeger JP, George KP, Hopman MT, Thijssen DH. Predictors of cardiac troponin release after a marathon. J Sci Med Sport. 2015 Jan;18(1):88-92. doi: 10.1016/j.jsams.2013.12.002. Epub 2014 Jan 2. PMID 24440407
- [Background] Serrano-Ostariz E, Legaz-Arrese A, Terreros-Blanco JL, Lopez-Ramon M, Cremades-Arroyos D, Carranza-Garcia LE, Izquierdo-Alvarez S, Bocos-Terraz P. Cardiac biomarkers and exercise duration and intensity during a cycle-touring event. Clin J Sport Med. 2009 Jul;19(4):293-9. doi: 10.1097/JSM.0b013e3181ab3c9d. PMID 19638823
- [Background] Eijsvogels T, George K, Shave R, Gaze D, Levine BD, Hopman MT, Thijssen DH. Effect of prolonged walking on cardiac troponin levels. Am J Cardiol. 2010 Jan 15;105(2):267-72. doi: 10.1016/j.amjcard.2009.08.679. PMID 20102930
- [Background] Neumayr G, Pfister R, Mitterbauer G, Maurer A, Gaenzer H, Sturm W, Hoertnagl H. Effect of the "Race Across The Alps" in elite cyclists on plasma cardiac troponins I and T. Am J Cardiol. 2002 Feb 15;89(4):484-6. doi: 10.1016/s0002-9149(01)02280-9. No abstract available. PMID 11835940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive sampling was done by voluntary confirmation of participants in the 2017 North Coast tour (http://ina-northcoast-cyclingtour.com/index.html) and the 2017 Tour de Borobudur (https://event.sambabikers.com/). All participants were invited to participate in this observational study via an online advertisement on the website.
Pre-assignment Details: Participants with a history of coronary artery diseases (CAD) were excluded from study participation. Subsequently, a total of 94 participants were included in this study
Groups:
- Group 140kms Cycling: willing to participate in 140kms cycling touring of TdB 2017
  140kms cycling: main exposure is long distance cycling touring (TdB/NC) consists of three groups; 140kms, 100kms and 240kms
- Group 100kms Cycling: willing to participate in 100kms cycling touring of TdB 2017
  140kms cycling: main exposure is long distance cycling touring (TdB/NC) consists of three groups; 140kms, 100kms and 240kms
- Group 240kms Cycling: willing to participate in 240kms cycling touring of NC 2017
  140kms cycling: main exposure is long distance cycling touring (TdB/NC) consists of three groups; 140kms, 100kms and 240kms
Period: Overall Study
Arm/Group | Group 140kms Cycling | Group 100kms Cycling | Group 240kms Cycling
Started | 32 | 34 | 28
Completed | 30 | 30 | 28
Not Completed | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Population: 30 participants completed Tour de Borobudur 140K, 2017 30 participants completed Tour de Borobudur 100K, 2017 28 participantas completed North Coast Tour, 2017
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 140kms Cycling | Group 100kms Cycling | Group 240kms Cycling | Total
Number analyzed (Participants) | 30 | 30 | 28 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 26 | 28 | 84
  >=65 years | 0 | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (9.33) | 43.5 (10.18) | 49.0 (13.70) | 45.3 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 30 | 30 | 28 | 88
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Indonesia | 30 | 30 | 28 | 88
cardiac troponin I (cTnI) [Mean (Standard Deviation); unit: ng/dL] | 5.2 (9.98) | 6.6 (10.56) | 3.5 (8.93) | 5.2 (9.83)

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Troponin I (cTnI)
Description: specific protein to determine cardiac injury
Time Frame: immediate after TdB 2017 cycling touring within less than 5 min
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Group 140kms Cycling | Group 100kms Cycling | Group 240kms Cycling
Number analyzed (Participants) | 30 | 30 | 28
ng/dL | 6.6 (46.6) | 10.1 (10.44) | 25.0 (61.39)

2. Primary Outcome: Malondialdehyde (MDA)
Description: oxydative stress marker
Time Frame: immediate after TdB 2017 cycling touring within less than 5 min
Measure: Mean (Standard Deviation); unit: mcmol/mL
Arm/Group | Group 140kms Cycling | Group 100kms Cycling | Group 240kms Cycling
Number analyzed (Participants) | 30 | 30 | 28
mcmol/mL | 206.1 (116.84) | 196.4 (68.59) | 231.2 (105.54)

3. Secondary Outcome: High Sensitivity C Reactive Protein (Hs-CRP)
Description: a biomarker that represents the inflammation process
Time Frame: immediate after TdB 2017 cycling touring within less than 5 min
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group 140kms Cycling | Group 100kms Cycling | Group 240kms Cycling
Number analyzed (Participants) | 30 | 30 | 28
mg/dL | 454 (286.5) | 335 (375.1) | 350 (332.6)

4. Secondary Outcome: Number of Participants With Pathological ECG Appearance
Description: Number of Participants with Pathological ECG Appearance.
  Pathological ECG appearance was the results of the ECG test describing one of the pathological appearances in ECG i.e.:
  1. The pathological rhythm which is may consist of Atrial Flutter, Atrial Fibrillation, Supraventricular Tachycardia, Ventricular Fibrillation, First Degree Heart Block, Second Degree Heart Block, Type 1 - Mobitz I, Second Degree Heart Block, Type 2 - Mobitz II, Third Degree Heart Block, or other pathological rhythm appearances
  2. Pathological ST-segment i.e. ST elevation (early repolarization), or another form
  3. Pathological U wave, and
  4. other pathological appearances
Time Frame: immediate after TdB 2017 cycling touring within less than 5 min
Population: Pathological ECG appearance
Measure: Count of Participants; unit: Participants
Arm/Group | Group 140kms Cycling | Group 100kms Cycling | Group 240kms Cycling
Number analyzed (Participants) | 30 | 30 | 28
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: during the event (cycling activity of TdB and NC) i.e. 6.1 hours range 3.5-9.8 and 24 hours after the event
Arm/Group | Group 140kms Cycling | Group 100kms Cycling | Group 240kms Cycling
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT03310450/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT03310450/SAP_001.pdf